CLINICAL TRIAL: NCT04250675
Title: Intermittent Pneumatic Compression to Improve the Outcome of Revascularization for Severe Peripheral Artery Disease: a Pilot Study
Brief Title: Intermittent Pneumatic Compression to Improve Revascularization Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Roseguini, Bruno, PhD (Individual)
Responsible Party: Principal Investigator, Raghu Motaganahalli, Associate Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1907961196
Record Dates: First submitted 2019-12-15; First posted 2020-01-31 (Actual); Results first posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Sham (Sham Comparator): Participants will apply Intermittent Pneumatic Compression (IPC) using a customized version of the Arterial Assist Device to both legs for 2 hours daily for a duration of 3 months. The sham device applies a compression sequence of 30 mmHg to the foot, ankle and calf with inflatable cuffs.
  Interventions: Device: Sham
- Active Comparator - Intermittent Pneumatic Compression (Active Comparator): Participants will apply Intermittent Pneumatic Compression (IPC) using the Arterial Assist Device to both legs for 2 hours daily for a duration of 3 months. The Arterial Assist Device® applies a compression sequence of 120 mmHg to the foot, ankle and calf with inflatable cuffs.
  Interventions: Device: Intermittent pneumatic leg compressions

INTERVENTIONS:
Device: Intermittent pneumatic leg compressions — Patients will be asked to use the ArtAssist® device to compress the foot and ankle (120 mmHg) of both legs for 2 hours daily for 3 months.
  Arms: Active Comparator - Intermittent Pneumatic Compression
Device: Sham — Patients will be asked to use the ArtAssist® device to compress the foot and ankle (30 mmHg) of both legs for 2 hours daily for 3 months.
  Arms: Sham

SUMMARY:
The purpose of this study is to investigate whether daily treatment with intermittent pneumatic leg compressions (IPC) following a nonsurgical vascular procedure improves circulation and enhances walking distance.

DETAILED DESCRIPTION:
Restenosis following revascularization procedures occur frequently and as early as 3 months after the intervention. There is an urgent need for adjunctive therapies that aid in the improvement of tissue blood flow and consequently relieve pain and improve functional capacity in these patients. It has been previously shown that exposure to IPC enhances leg blood flow to collateral-dependent tissues. In this study, subjects who have undergone nonsurgical revascularization will be randomly assigned to two groups: IPC or placebo pump. Subjects will receive a commercially available IPC device (Art Assist, ACI Medical, San Marcos, CA) and will apply the treatment at home for 2 hours daily over 3 consecutive months. At 3 time points (pre, 1 and 3 months post procedure) assessments will be performed (hemodynamics, rest pain, calf muscle oxygenation during exercise, walking endurance and quality of life).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Scheduled for endovascular revascularization of one or both lower extremities.

Exclusion Criteria:

* Chronic kidney disease (eGFR <30 by MDRD or Mayo or Cockcroft-Gault formula)
* Open and/or non-healing wounds in the areas covered by IPC cuff
* Walking limited by a symptom other than PAD
* Presence of any clinical condition that makes the patient unsuitable to participate in the trial
* Concern for inability of the patient to comply with study procedures and/or follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- IU Health Methodist, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sham | Active Comparator - Intermittent Pneumatic Compression
Started | 5 | 4
Completed | 4 | 4
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham | Active Comparator - Intermittent Pneumatic Compression | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 3 | 2 | 5
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68 (8) | 62 (6) | 66 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 2 | 4 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 4 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Walking Endurance
Description: Change in 6 Minute Walk Test from baseline to 3 months
Time Frame: Baseline and after 1 and 3 months of treatment
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Sham | Active Comparator - Intermittent Pneumatic Compression
Number analyzed (Participants) | 4 | 4
Meters | -14 (25) | 35 (38)

2. Secondary Outcome: Ankle-brachial Index (ABI)
Description: Change in ABI from baseline to 3 months. A handheld 5-MHz Doppler ultrasound (Lumeon, McKesson) was used to obtain duplicate measurements of systolic pressures in the right posterior tibial artery, right dorsalis pedis artery, right brachial artery, left posterior tibial artery, left dorsalis pedis artery, and left brachial artery. The ABI of each leg was calculated by dividing the higher of the dorsalis pedis pressure or posterior tibial pressure by the higher of the right or left arm blood pressure
Time Frame: Baseline and after 3 months of treatment
Measure: Mean (Standard Deviation); unit: AU
Arm/Group | Sham | Active Comparator - Intermittent Pneumatic Compression
Number analyzed (Participants) | 4 | 4
AU | 0.04 (0.07) | -0.03 (0.07)

3. Secondary Outcome: Vascular Quality of Life Score (VascuQol)
Description: Change in scores for VascuQol Questionnaire from baseline to 3 months. Overall score range is 7-175; higher score means higher quality of life.
Time Frame: Baseline and after 1 and 3 months treatment
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Sham | Active Comparator - Intermittent Pneumatic Compression
Number analyzed (Participants) | 4 | 4
Units on a scale | 0.07 (0.34) | 0.22 (0.67)

4. Secondary Outcome: Toe-brachial Index
Description: Change in toe-brachial index from baseline to 3 months. A toe-brachial index (TBI) is a non-invasive test that measures the ratio of systolic blood pressure in the toe to the higher systolic pressure in the arm. A toe/digit pressure cuff is wrapped around the measured toe, and a senso is placed on the toe distally to the pressure cuff.
Time Frame: Baseline and after 1 and 3 months of treatment
Measure: Mean (Standard Deviation); unit: U
Arm/Group | Sham | Active Comparator - Intermittent Pneumatic Compression
Number analyzed (Participants) | 4 | 4
U | 0.04 (0.19) | -0.03 (0.07)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Sham | Active Comparator - Intermittent Pneumatic Compression
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/4
Other Adverse Events (participants affected / at risk) | 1/5 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham (N=5) | Active Comparator - Intermittent Pneumatic Compression (N=4)
Hyperkalemia (Blood and lymphatic system disorders) | 0 | 1 (1) — Baseline lab results drawn showed an elevated serum potassium (6.5 mmol/L).
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham (N=5) | Active Comparator - Intermittent Pneumatic Compression (N=4)
Leg discomfort during treatment (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Leg discomfort during treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-29): https://cdn.clinicaltrials.gov/large-docs/75/NCT04250675/Prot_SAP_001.pdf